CLINICAL TRIAL: NCT07406308
Title: A Comparative Analysis of Mid- to Long-Term Outcomes of Paclitaxel-Coated Balloon Angioplasty With Adjunctive Debulking Versus Paclitaxel-Coated Balloon Angioplasty Alone for the Treatment of Chronic Femoropopliteal Artery Occlusions
Brief Title: A Comparative Analysis of Mid- to Long-Term Outcomes: Paclitaxel-Coated Balloon With Debulking Versus Paclitaxel-Coated Balloon Alone in the Treatment of Chronic Femoropopliteal Artery Occlusions
Acronym: DCB-Debulk-COM
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCB_ATH
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Femoropopliteal Artery Occlusion
Keywords: Femoropopliteal Artery Occlusion; Drug-Coated Balloon; debulking procedures

STUDY DESIGN:
Intervention Model Description: This is a prospective, non-randomized, controlled cohort study.
  1. Eligible patients with chronic femoropopliteal artery occlusions will be assigned to one of the two treatment groups based on a combination of clinical assessment, anatomical factors, and patient preference: (1) the Combination Therapy Group (paclitaxel-coated balloon angioplasty with adjunctive atherectomy/debulking), or (2) the DCB-Alone Group (paclitaxel-coated balloon angioplasty alone).
  2. Treatment allocation is not randomized. Patients in both groups will be prospectively followed and their outcomes compared to assess the relative efficacy and safety of the two treatment strategies.
Masking Description: Masking Description
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB (Active Comparator): Participants in this group will be received drug-coated balloon angioplasty
  Interventions: Device: paclitaxel-coated balloon angioplasty
- DCB+DP (Experimental): Participants in this group will be received drug-coated balloon angioplasty with debulking procedures.
  Interventions: Device: paclitaxel-coated balloon angioplasty with debulking procedures

INTERVENTIONS:
Device: paclitaxel-coated balloon angioplasty — No debulking procedures were taken
  Arms: DCB
Device: paclitaxel-coated balloon angioplasty with debulking procedures — The patient underwent DCB treatment along with debulking procedures (such as laser or plaque rotational atherectomy, etc.).
  Arms: DCB+DP

SUMMARY:
This study aims to compare mid-to long-term outcomes of paclitaxel-coated balloon angioplasty with adjunctive debulking versus paclitaxel-coated balloon angioplasty alone for the treatment of chronic femoropopliteal artery diseases.

DETAILED DESCRIPTION:
Chronic femoropopliteal artery occlusion, particularly in long lesions, remains a significant challenge in endovascular treatment of lower extremity arterial disease due to its high occlusion burden and severe vascular calcification. In recent years, with the continuous advancement of endovascular techniques and devices, especially the emergence of the "leave nothing behind" concept, Drug-Coated Balloon (DCB) angioplasty has become a mainstream approach for treating femoropopliteal occlusions. While DCB offers excellent long-term patency and preserves future treatment options, adjunctive debulking procedures-a category of techniques that physically remove or ablate plaque prior to DCB dilation to achieve a larger, smoother lumen-have gained attention. These techniques primarily include atherectomy, laser ablation, and directional atherectomy. They can address more complex lesions and offer potential benefits such as enhanced drug absorption, reduced elastic recoil, and decreased need for bailout stenting. However, they also carry risks, including distal embolism and perforation. Consequently, the comparative efficacy between DCB alone and DCB combined with debulking measures remains uncertain, and the choice of treatment strategy still largely depends on operator experience. Therefore, an in-depth investigation is necessary to compare the efficacy and safety of these two approaches to inform and guide optimal clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Subject age 18-85yrs.
* Subject has been informed of the nature of the study, agrees to participate, and has signed a Medical Ethics Committee approved consent form.
* Subject understands the duration of the study, agrees to attend follow-up visits, and agrees to complete the required testing.
* Rutherford category 2-5.
* Subject has atherosclerotic de novo, non-stented restenotic, or in-stent restenotic/occlusive lesions in the superficial femoral artery (SFA) and/or popliteal artery (P1 segment).
* Patent inflow artery with stenosis <30% by visual estimation (or by core lab assessment if available) and at least 1 infrapopliteal artery to the ankle (<50% diameter stenosis).
* A guidewire has successfully traversed the target treatment segment.

Exclusion Criteria:

* Subject presents with acute arterial embolism or thrombosis requiring thrombectomy or thrombolysis for limb ischemia.
* Subject has arterial occlusion caused by thromboangiitis obliterans (Buerger's disease) or other forms of immune-mediated vasculitis.
* Subject has undergone surgery on the target vessel within the past 3 months, or has experienced repeated failures of endovascular therapy and is deemed unsuitable for further endovascular intervention.
* Subject has an uncontrolled thrombophilia or hypercoagulable state.
* Subject has a severe systemic disease (e.g., malignancy) with a life expectancy of less than 1 year.
* Subject has contraindications or intolerance to antiplatelet/anticoagulant medications, such as aspirin, clopidogrel, or heparin.
* Subject is pregnant or breastfeeding.
* Subject meets one or more of the following conditions: chronic renal insufficiency (SCr ≥ 2.5 mg/dL) or on regular dialysis; cardiovascular or cerebrovascular surgery within the past 1 month; or severe sequelae from a major stroke.
* Subject has a known allergy to nitinol alloy, paclitaxel, or contrast agents.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2026-04-20 (Estimated); Primary Completion 2028-03-20 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
1-year primary patency rate | 1 year

SECONDARY OUTCOMES:
free from clinical-driven target lesion revascularization | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided